CLINICAL TRIAL: NCT05664620
Title: Development of a Persisting Concussion Symptoms (PCS) Risk Stratification Tool and Evaluation of the Effectiveness of an Enhanced WSIB Multidisciplinary Individualized Treatment Program to Enhance Return to Work and Recovery
Brief Title: Post Concussion Symptoms Risk Stratification Tool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-6079
Record Dates: First submitted 2022-11-22; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Post-Concussion Syndrome
MeSH Terms: conditions — Post-Concussion Syndrome

STUDY DESIGN:
Intervention Model Description: Diagnostic Test: Risk Stratification Tool Patients will be allocated to three groups (Low, medium and high risk) by using the Risk Stratification Tool, and High-risk patients will receive multidisciplinary treatment assigned to them by a physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low risk (No Intervention): Standard of care to treat post-concussion symptoms in the community
- Medium risk (No Intervention): Patients who are assigned to the medium risk group will receive the same treatment as the low risk group for one month, after which they will be reassessed. If improving they will go into the low risk group, and if not improving they will go into the high risk group
- High risk (Other): A multidisciplinary individualized treatment (personalized medicine) model of treating all post-concussion symptoms simultaneously including the following:
  Headache therapy, balance therapy, vestibular therapy, exercise therapy* mental health support e.g. CBT and/or mindfulness meditation* (with more specialized diagnosis and care where required), cognitive assessment and therapy, vision therapy, sleep assessment and therapy, physiotherapy, education sessions*, occupational therapy These patients will be treated through the Altum Health Neurology Specialty Program
  *Offered to all high risk patients
  Interventions: Diagnostic Test: Risk Stratification Tool

INTERVENTIONS:
Diagnostic Test: Risk Stratification Tool — Patients will be allocated to three groups (Low,medium and high risk) by using the Risk Stratification Tool, and High risk patients will receive multidisciplinary treatment assigned to them by a physician
  Arms: High risk

SUMMARY:
Patients with Persisting Concussion Symptoms (PCS) have a multitude of different symptoms. Some patients are at risk of prolonged symptoms but currently there is no tool to assist in identifying patients at high risk. Intensive, multidisciplinary intervention is time-consuming and expensive and may not be warranted for all PCS patients, so it is essential to identify early on which patients are at risk of prolonged symptoms. The aim of this study is to improve the quality of care delivered to patients, especially those who are at high-risk of prolonged PCS by early identification and treatment of all the symptoms. The purpose of this research is to validate the use of a Persisting Concussion Symptoms (PCS) Risk Stratification Tool (RST).

DETAILED DESCRIPTION:
The information from 500 hundred concussion patients were used to develop the PCS RST. This is a screening tool that will assist in predicting patient outcomes by allocating patients with PCS into a low, medium and high risk group for prolonged PCS symptoms. This categorization would help target those patients at high risk of prolonged symptoms with a multidisciplinary individualized treatment and evaluate the effectiveness of it on return to work and recovery. For this research study, we ask workers who have had concussions and are categorized as high high risk (with PCS RST) for prolonged PCS symptoms to undergo individualized treatments and we will examine their recovery and return to work.

The study will involve 75 patients with persisting concussion symptoms from the Canadian Concussion Centre clinics and Altum Health concussion clinic at Toronto Western Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-60 years old
2. Clinical diagnosis of PCS for 1-12 months with at least 3 symptoms
3. Must be employed at time of injury
4. Full-time or part-time worker prior to concussion and cannot return to work
5. Must speak English and be sufficiently literate to complete questionnaires and perform assessments
6. Must be able to give consent

Exclusion Criteria:

1. Abnormalities on MRI such as contusion, hemorrhages, siderosis, or other non-traumatic conditions
2. History of neurological conditions (e.g. stroke, seizures) or major psychiatric disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Return to work | 12 months after treatment start day
  The Primary Outcome is the percentage of concussed workers who ultimately RTW one year after the treatment commences. The Recovery and Return to Work tracker will be completed in 3,6,9 and 12 months to track their recovery. However, the primary endpoint is "Return to work at 12 months."

SECONDARY OUTCOMES:
Work Quality | 12 months after treatment start day
  The type of work returned to in relation to the pre-concussion work and work stability in terms of being able to stay working after RTW. For this purpose, a modified work quality Index (WQI) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Tator, MD, PhD, Principal Investigator — University Health Network, Toronto; Carmela Tartaglia, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Canadian Concussion Centre- Toronto Western Hospital, Toronto, Ontario, Canada